CLINICAL TRIAL: NCT01357512
Title: Evaluation of Diagnostic Value of 3-T MRI in Suspected Prostate Cancer
Brief Title: Evaluation of Diagnostic Value of 3-T Magnetic Resonance Imaging (MRI) in Suspected Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Markku Vaarala, MD, PhD, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRODIAMRI
Record Dates: First submitted 2011-04-14; First posted 2011-05-20 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer diagnosis; magnetic resonance imaging; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI done (Experimental): Subjects with MRI prior prostate biopsies
  Interventions: Device: magnetic resonance imaging, Siemens
- no MRI (No Intervention): No MRI before prostate biopsies

INTERVENTIONS:
Device: magnetic resonance imaging, Siemens — Magnetic resonance imaging (MRI) of prostate with Siemens 3-tesla device
  Arms: MRI done

SUMMARY:
The purpose of the study is to evaluate the usefulness of 3-T magnetic resonance imaging (MRI) in the evaluation of suspected prostate cancer. Men with suspected prostate cancer based on serum prostate-specific antigen antigen (PSA) value are included. Men are randomized to pre-biopsy MRI or no MRI groups in ratio 1:1. Standard transrectal ultrasound guided biopsies will be taken in addition to extra biopsies from lesions suspicious based on MRI evaluation. Hypothesis is that more prostate cancers will be found after MRI evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Suspected prostate cancer based on PSA value (total PSA 2,5-10 ng/ml and PSA free to total ratio <=0.15, or total PSA 10-20 ng/ml)
* PSA and serum creatinine measurement less than 60 days before transrectal ultrasound-guided prostate biopsies
* No evidence of PSA increase by non-cancerous factors (catheterization, bladder stones, urinary tract infection including bacterial prostatitis)

Exclusion Criteria:

* Previous prostate biopsies
* Previous prostate surgery
* Contraindication for MRI (such as pacemaker or inner ear implant)
* Claustrophobia
* Estimated glomerular filtration rate (eGFR) <40 ml/min
* Suspected clinical T3-T4 prostate cancer based on digital rectal examination
* Contraindication for transrectal ultrasound-guided prostate biopsies
* body mass index >30

Ages: 40 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markku Vaarala, MD PhD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Tonttila PP, Lantto J, Paakko E, Piippo U, Kauppila S, Lammentausta E, Ohtonen P, Vaarala MH. Prebiopsy Multiparametric Magnetic Resonance Imaging for Prostate Cancer Diagnosis in Biopsy-naive Men with Suspected Prostate Cancer Based on Elevated Prostate-specific Antigen Values: Results from a Randomized Prospective Blinded Controlled Trial. Eur Urol. 2016 Mar;69(3):419-25. doi: 10.1016/j.eururo.2015.05.024. Epub 2015 May 29. PMID 26033153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI Done | no MRI
Started | 65 | 65
Completed | 53 | 60
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Population: Population with protocol violations excluded
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI Done | no MRI | Total
Number analyzed (Participants) | 53 | 60 | 113
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [60 to 66] | 62 [56 to 67] | 62 [58 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 60 | 113
Region of Enrollment [Number; unit: participants]
  Finland | 53 | 60 | 113
Serum prostate-specific antigen level [Median (Inter-Quartile Range); unit: ng/ml] | 6.1 [4.2 to 9.9] | 6.2 [4.0 to 10.7] | 6.1 [4.1 to 10.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Prostate Cancer Diagnoses in MRI and no MRI Groups
Description: The number of patients with confirmed prostate cancer among men with MRI performed before biopsies are compared to the number of patients with prostate cancer confirmed in prostate biopsies without MRI. The number patients with prostate cancer are counted as total from cancers detected in random biopsies and in biopsies targeted based on suspicious MRI findings in MRI group, and from random biopsies in no MRI group.
Time Frame: at the end of the study (up to 1 year)
Measure: Number; unit: participants
Arm/Group | MRI Done | no MRI
Number analyzed (Participants) | 53 | 60
participants | 34 | 34

2. Secondary Outcome: Number of Positive Biopsies in MRI and no MRI Groups
Description: The number of biopsies with histology confirming prostate cancer are compared between MRI and no MRI groups. This measure will clarify if prostate cancer can be diagnosed more accurately, i.e. more biopsies with confirmed prostate cancer, after MRI. Ten or 12 biopsies will be taken from prostates below 30 grams, or equal or above 30 grams, respectively.
Time Frame: at the end of the study (up to 1 year)
Measure: Median (Inter-Quartile Range); unit: number of cancer-positive biopsy cores
Arm/Group | MRI Done | no MRI
Number analyzed (Participants) | 53 | 60
number of cancer-positive biopsy cores | 3.0 [2.0 to 5.0] | 3.0 [1.75 to 5.25]

3. Secondary Outcome: Proportion of Clinically Significant Prostate Cancers Detected in MRI and no MRI Groups
Description: Number of clinically significant prostate cancers detected with and without MRI. Clinically significant prostate cancer is determined by the Gleason grading and be the number of cancer-positive biopsy cores.
Time Frame: at the end of the study (up to 1 year)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | MRI Done | no MRI
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/60
Other Adverse Events (participants affected / at risk) | 0/53 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Done (N=53) | no MRI (N=60)
collapse (Cardiac disorders) | 0 (0) | 1 (1) — Collapse after prostate biopsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No